CLINICAL TRIAL: NCT07229430
Title: A Prospective, Multi-center, Randomized Controlled, Non-inferiority Study to Evaluate the Safety and Effectiveness of ULTRAFORMER MPT PLUS Treatment to Lift Lax Submental (Beneath the Chin) and Neck Tissue
Brief Title: Safety and Effectiveness Evaluation of the High-intensity Focused Ultrasound Device for Lifting Lax Submental and Neck Tissue
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: CLASSYS Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CS-483
Record Dates: First submitted 2025-11-13; First posted 2025-11-17 (Actual); Last update posted 2025-12-01 (Actual); Status verified 2025-11

CONDITIONS: Skin Laxity (Submental and Neck); Facial Skin Laxity; Submental Tissue Laxity
Keywords: ULTRAFORMER MPT PLUS; High-Intensity Focused Ultrasound; HIFU; Submental Lifting; Skin Laxity; Non-surgical Lift; Aesthetic Device; Classys; Non-Inferiority Clinical Trial
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to receive either ULTRAFORMER MPT PLUS treatment or the comparator device (Ulthera® System). Each subject receives a single assigned treatment without crossover.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study is evaluator-blinded. Participants and outcomes assessors will remain blinded to treatment allocation, while treatment providers will be unblinded to operate the assigned device.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- ULTRAFORMER MPT PLUS Group (Experimental): ULTRAFORMER MPT PLUS (Classys Inc., Seoul, Korea) delivers high-intensity focused ultrasound (HIFU) energy to the subdermal tissue to induce neocollagenesis and tissue contraction for non-surgical skin tightening and lifting.
  Interventions: Device: ULTRAFORMER MPT PLUS
- Ulthera Comparator Group (Active Comparator): The Ulthera® System (Merz Aesthetics, USA) uses focused ultrasound energy to lift and tighten submental and neck skin and serves as the reference comparator in this non-inferiority clinical trial.
  Interventions: Device: Ulthera System

INTERVENTIONS:
Device: ULTRAFORMER MPT PLUS — ULTRAFORMER MPT PLUS (Classys Inc., Seoul, Korea) is a high-intensity focused ultrasound (HIFU) system that delivers focused energy at multiple depths to induce neocollagenesis and tissue contraction for non-surgical lifting and tightening of submental and neck tissue. The device includes both Default and MP modes and is under investigation under FDA IDE G250041.
  Arms: ULTRAFORMER MPT PLUS Group
Device: Ulthera System — The Ulthera System (Merz Aesthetics, USA) is an FDA-cleared high-intensity focused ultrasound (HIFU) device indicated for non-invasive lifting and tightening of lax tissue in the submental and neck areas. It serves as the active comparator for this non-inferiority clinical study.
  Arms: Ulthera Comparator Group

SUMMARY:
This is a prospective, multicenter, randomized, evaluator-blinded, parallel-controlled, non-inferiority clinical study designed to evaluate the safety and effectiveness of the ULTRAFORMER MPT PLUS, a high-intensity focused ultrasound (HIFU) device, for lifting and tightening lax submental (beneath the chin) and neck tissue in adult subjects.

Approximately 273 subjects will be enrolled at multiple investigational sites across the United States.

Participants will receive either the ULTRAFORMER MPT PLUS treatment or the predicate comparator device, and will be followed for safety and efficacy assessments including clinical photography, investigator evaluation, and patient-reported outcomes.

The study aims to demonstrate that ULTRAFORMER MPT PLUS is non-inferior to the approved reference device in improving skin laxity and wrinkle appearance of the lower face and neck.

DETAILED DESCRIPTION:
This prospective, multicenter, randomized, evaluator-blinded, parallel-controlled, non-inferiority clinical investigation is conducted under an FDA Investigational Device Exemption (IDE #G250041) to evaluate the safety and effectiveness of the ULTRAFORMER MPT PLUS (Class II high-intensity focused ultrasound system) for aesthetic improvement of submental and neck tissue laxity.

A total of approximately 273 subjects aged 30-65 years with mild-to-moderate skin laxity in the submental and neck areas will be enrolled across up to 5 U.S. investigational sites. Subjects will be randomized 1:1 to receive either ULTRAFORMER MPT PLUS or the comparator device (ULTHERA® System, Merz Aesthetics, USA).

Primary endpoints include blinded investigator-assessed improvement using the validated Facial Laxity Grading Scale and safety outcomes based on the incidence and severity of device-related adverse events. Secondary endpoints include participant-reported improvement scores, digital image analysis, and durability of effect at 8-week and 12-week follow-ups.

The study consists of two sequential safety stages (Stage 1A and 1B; 20 subjects total) followed by the pivotal Stage 2 phase (approximately 253 subjects). Data from the safety stages will be reviewed by an independent Data Safety Monitoring Board (DSMB) prior to progression to Stage 2.

All treatments will be performed by trained investigators according to the protocol-defined parameters. Subjects will be evaluated at baseline, post-treatment, and during follow-up visits up to 6 months. The final statistical analysis will assess non-inferiority of ULTRAFORMER MPT PLUS to the predicate device with respect to the primary efficacy endpoint and confirm overall safety.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 30 to 65 years, inclusive, at the time of informed consent.
2. Subjects presenting with mild to moderate submental and/or neck skin laxity, as determined by the investigator.
3. Subjects in good general health with stable body weight (±5%) for at least 6 months prior to screening.
4. Subjects willing to avoid other aesthetic or dermatologic procedures (surgical or non-surgical) to the treatment area during the study period.
5. Subjects able to understand and sign informed consent and comply with all study visits and procedures.
6. Female subjects of child-bearing potential who agree to use reliable contraception throughout study participation.

Exclusion Criteria:

1. Prior facelift, neck lift, liposuction, or contouring surgery involving the lower face, submental, or neck areas.
2. Receipt of any energy-based aesthetic treatment (e.g., HIFU, radiofrequency, laser) or injectable aesthetic treatment (e.g., botulinum toxin, dermal filler, collagen stimulator) to the treatment area within 6 months prior to baseline.
3. Presence of any implanted electronic medical device, such as a pacemaker, defibrillator, or neurostimulator.
4. Active skin infection, wound, cystic acne, inflammation, or severe scarring within or near the treatment area.
5. History of keloid formation or abnormal wound healing.
6. Known bleeding disorder, or use of anticoagulant or antiplatelet medications that cannot be safely discontinued for the procedure.
7. Pregnant or breastfeeding women.
8. Subjects with a known sensitivity or contraindication to ultrasound-based procedures.
9. Any medical or psychiatric condition that, in the investigator's judgment, could interfere with study participation, safety, or data integrity.
10. Participation in another investigational study within 30 days prior to screening.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 273 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2026-11-26 (Estimated); Study Completion 2026-11-26 (Estimated)

PRIMARY OUTCOMES:
Submental Area Lift [Time Frame: 90 Days Post-Treatment] | 90 Days Post-Treatment
  The primary endpoint of the study is the Submental Area Lift "Success" evaluated at 90 days post-treatment.
  A "Success" is defined as a reduction in the measured submental area of ≥ 20 mm² compared with baseline. Both left and right lateral 2D images will be derived from 3D photographs and analyzed by certified technicians using the Submental Lift Application (Canfield Scientific Inc.).

SECONDARY OUTCOMES:
Submental Area Lift [Time Frame: 60 Days Post-Treatment] | 60 Days Post-Treatment
  Submental Area Lift ≥ 20 mm² vs baseline.
Submental Area Lift [Time Frame: 90 Days Post-Treatment] | 90 Days Post-Treatment
  Submental Area Lift ≥ 20 mm² vs baseline.
Change in Overall Lifting of Treated Tissue on Submental and Neck Regions [Time Frame: 60 and 90 Days Post-Treatment] | 60 and 90 Days Post-Treatment
  Percentage of patients assessed to have improvement in skin laxity (lifted skin) by ≥ 2 of 3 independent blinded evaluators comparing pre-, 60-, and 90-day post-treatment images. Images will be prepared and randomized for review per Canfield SOPs (FDA K121700).
Global Aesthetic Improvement Scale (GAIS) Results [Time Frame: 60 and 90 Days Post-Treatment] | 60 and 90 Days Post-Treatment
  Overall aesthetic improvement rated on a 5-point scale (1 = Very Much Improved to 5 = Worse) by the investigator comparing pre- and post-treatment photographs. Assessed by PI or delegated qualified staff at each visit.
Subject Satisfaction Questionnaire[Time Frame: 60 and 90 Days Post-Treatment] | 60 and 90 Days Post-Treatment
  5-point Likert scale (1 = Very Satisfied to 5 = Very Dissatisfied). "Satisfied" = Very Satisfied or Satisfied.
  Completed at each follow-up visit.
Visual Analog Scale (VAS) - Pain Score[Time Frame:Immediately Post-Treatment] | Immediately Post-Treatment
  Subject-reported pain (0 = No pain, 10 = Worst pain possible) recorded immediately after treatment completion.
  Pain management at investigator's discretion; if applicable, documented as AE.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Rebecca Fitzgerald, MD, Inc., Los Angeles, California
  - Dermatology, Laser & Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Wilmington Dermatology Center, Wilmington, North Carolina
  - Nashville Centre for Laser and Facial Surgery, Nashville, Tennessee
  - Spokane Dermatology Clinic / Werschler Aesthetics, Spokane, Washington

IPD SHARING:
Plan to Share IPD: No